CLINICAL TRIAL: NCT04907968
Title: Upifitamab Rilsodotin (Xmt-1536) An Open-Label, Multicenter, Dose Escalation And Expansion Study Of Upifitamab Rilsodotin In Combination With Carboplatin In Participants With High Grade Serous Ovarian Cancer (Upgrade-A)
Brief Title: Study of Upifitamab Rilsodotin in Combination With Carboplatin in Participants With High-grade Serous Ovarian Cancer
Acronym: UPGRADE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Terminated by Sponsor
Sponsor: Mersana Therapeutics (Industry)
Collaborators: IQVIA Biotech (Industry); PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMT-1536-2A
Record Dates: First submitted 2021-05-12; First posted 2021-06-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Platinum-sensitive Ovarian Cancer (UPGRADE-A)
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation - Module A (UPGRADE-A) (Experimental): XMT-1536 (Upifitabmab Rilsodotin) + carboplatin is administered in groups of patients who will receive doses of XMT-1536 that increase over time.
  Interventions: Drug: XMT-1536 (Upifitamab Rilsodotin); Drug: Carboplatin
- Dose Expansion - Module A (UPGRADE-A) (Experimental): Once the MTD or RP2D is achieved in dose escalation, a new group of patients will receive XMT-1536 (Upifitamab Rilsodotin) at this fixed-dose + carboplatin.
  Interventions: Drug: XMT-1536 (Upifitamab Rilsodotin); Drug: Carboplatin

INTERVENTIONS:
Drug: XMT-1536 (Upifitamab Rilsodotin) — Drug: XMT-1536 (Upifitamab Rilsodotin) XMT-1536 (Upifitamab Rilsodotin) will be administered on Day 1 of each 28-day cycle until disease progression, unacceptable toxicity, or either the patient or study physician determines it is in the best interest of the patient to discontinue participation in the study
  Other Names:
  * XMT-1536
  * UpRi Drug: Carboplatin Carboplatin will be administered on Day 1 on each of the first six 28 day cycles.
  Other Names: XMT-1536; UpRi
Drug: Carboplatin — Drug: XMT-1536 (Upifitamab Rilsodotin) XMT-1536 (Upifitamab Rilsodotin) will be administered on Day 1 of each 28-day cycle until disease progression, unacceptable toxicity, or either the patient or study physician determines it is in the best interest of the patient to discontinue participation in the study
  Other Names:
  * XMT-1536
  * UpRi Drug: Carboplatin Carboplatin will be administered on Day 1 on each of the first six 28 day cycles.

SUMMARY:
Phase 1 safety study of the antibody-drug conjugate (ADC) XMT-1536 (upifitamab rilsodotin) administered as an intravenous infusion once every four weeks in combination with Carboplatin in participants with high-grade serous ovarian cancer (HGSOC, including fallopian tube and primary peritoneal cancer). The trial consists of dose escalation (DES) and expansion (EXP) portion. In addition to safety assessments, the pharmacokinetics of the drug will be assessed along with ADC activity.

DETAILED DESCRIPTION:
This trial is an open-label, multi-center Phase 1 study of upifitamab rilsodotin administered as an intravenous infusion once every 28 days in combination with Carboplatinin patients with high-grade serous ovarian cancer (HGSOC, including fallopian tube and primary peritoneal cancer). The trial consists of dose escalation (DES) and expansion (EXP) portion. The primary objective of the dose escalation (DES) portion is to establish the maximum tolerated dose (MTD) for upifitamab rilsodotin in combination with Carboplatin. In the EXP portion of the trial, participants will initiate treatment at the MTD or recommended phase 2 dose (RP2D) determined in the DES for the combination.

ELIGIBILITY:
Inclusion Criteria:

Participant must be at least 18 years of age, and female; Participant must be able to understand the study procedures and agree to participate in the study by providing informed consent

* Participants must have a histological diagnosis of metastatic or recurrent high-grade serous ovarian cancer, which includes fallopian tube, or primary peritoneal cancer.
* Participant has received 1 to 3 prior lines of therapy for their ovarian cancer; a non-platinum-based chemotherapy regimen is permitted provided it is not the most recent line of therapy. Participant must have platinum-sensitive recurrent disease
* Participant must have an ECOG performance status 0 or 1
* Participant must have measurable disease as per RECIST v1.1
* Tumor sample must be provided, either an archival tumor tissue block or slides or, if not available, a tumor tissue block or slides from a new tumor biopsy obtained through a low-risk, medically routine procedure.
* Participants with toxicity from prior therapy or surgical procedures must have recovered to ≤ Grade 1. Participants with alopecia, stable immune-related toxicity such as hypothyroidism on hormone replacement, or adrenal insufficiency treated with ≤10 mg daily prednisone (or equivalent), after prior taxane therapy are exceptions to this criterion and may qualify for this study.
* Participants must have cardiac left ventricular ejection fraction (LVEF) ≥50% or ≥ the institution's lower limit of normal as measured by either Echo or MUGA scan
* Participants must have adequate organ function within 14 days prior to enrollment
* A female participant is eligible to participate if she is not pregnant or breastfeeding, if she is not a woman of childbearing potential (WOCBP), or if she is a WOCBP potential and using a contraceptive method that is highly effective.

Exclusion Criteria:

* Participant has known sensitivity to any of the study medications, or components thereof, or a history of drug or allergy that contraindicates their participation
* Participant is unable or unlikely to comply with dosing schedule and study evaluations.
* Participant has a prior hypersensitivity reaction to carboplatin requiring desensitization or discontinuation.
* Participant has prior platelet or neutrophil toxicity to carboplatin-containing therapy requiring dose reduction to AUC <5 mg x mL/min in the most recent regimen containing carboplatin
* Known history of CTCAE version 5.0 Grade 4 thrombocytopenia OR history of bleeding in association with any grade thrombocytopenia
* Participant has had major surgery within 28 days of starting study treatment, systemic anticancer therapy within the lesser of 28 days or 5 half-lives of the prior therapy before starting study treatment (14 days or 5 half-lives for small molecule targeted therapy), or recent radiation therapy with unresolved toxicity or within a time window of potential toxicity
* Participant has received prior treatment with mirvetuximab soravtansine or another ADC containing an auristatin or maytansinoid payload.
* Participant has untreated CNS metastases (including new and progressive brain metastases), history of leptomeningeal metastasis, or carcinomatous meningitis.
* Has a diagnosis of additional malignancy that required treatment within 2 years prior to screening, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix
* Participant is unwilling to be transfused with blood components.
* Participant is receiving concurrent anti-cancer therapy (e.g. chemotherapy, radiation therapy, biologic therapy, immunotherapy, hormonal therapy, investigational therapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
DES: Maximum tolerated dose (MTD) for Upifitamab Rilsodotin with carboplatin | Up to 24 weeks, from the date of first dose until unacceptable side effects or a dose-limiting toxicity is met
  Determine the MTD of Upifitamab rilsodotin in combination with carboplatin by evaluating adverse events in combination with carboplatin
EXP: Assess the feasibility of Upifitamab rilsodotin combination initiated at MTD or RP2D | First dose up until 30 days after study termination
  Assess the feasibility of Upifitamab rilsodotin combination initiated at MTD or RP2D Assess the feasibility of Upifitamab rilsodotin combination initiated at MTD or RP2D, where the regimen will be considered feasible if at least 60% of participants complete at least four cycles of the carboplatin-upifitamab rilsodotin combination, allowing for standard treatment modifications, without discontinuing treatment earlier for reasons other than disease progression

SECONDARY OUTCOMES:
DES and EXP: Safety and Tolerability, by observance of frequency and grade of adverse events based on CTCAE v5.0. | First dose up until 30 days after study termination
  DES and EXP: Safety and Tolerability, by observance of frequency and grade of adverse events based on CTCAE v5.0.
DES and EXP: Time of maximum observed concentration of carboplatin | Daily for one week after first dose; weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent
  Determine the pharmacokinetics of carboplatin
DES and EXP: Maximum concentration of XMT-1536 (Upifitamab rilsodotin) | weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1536 (Upifitamab rilsodotin)
DES and EXP: Maximum concentration of carboplatin | Weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of carboplatin
DES and EXP: Area under the concentration curve of the last measurable concentration of XMT-1536 (upifitamab rilsodotin) | Weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1536 (Upifitamab rilsodotin)
DES and EXP: Area under the concentration curve of the last measurable concentration of carboplatin | Weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of carboplatin
DES and EXP: Anti-neoplastic effects of XMT-1536 (Upifitamab rilsodotin) in combination with carboplatin | Every 8 weeks for the first 12 months, then every 12 weeks on treatment
  ORR (by RECIST 1.1)
DES and EXP: Anti-neoplastic effects of XMT-1536 (Upifitamab rilsodotin) in combination with carboplatin | Every 8 weeks for the first 12 months, then every 12 weeks on treatment
  DOR
DES and EXP: Anti-neoplastic effects of XMT-1536 (Upifitamab rilsodotin) in combination with carboplatin | Every 8 weeks for the first 12 months, then every 12 weeks on treatment
  DCR
DES and EXP: Anti-neoplastic effects of XMT-1536 (Upifitamab rilsodotin) in combination with carboplatin PFS (by RECIST 1.1) | Every 8 weeks for the first 12 months, then every 12 weeks on treatment
  PFS (by RECIST 1.1)
DES and EXP: Anti-neoplastic effects of XMT-1536 (Upifitamab rilsodotin) in combination with carboplatin | Every 90 days
  OS
DES and EXP: Assess the correlation of tumor expression of NaPi2b and objective tumor response | Every 8 weeks for the first 12 months, every 12 weeks on treatment, every 90 days for OS
  Potential NaPi2b protein or RNA levels of NaPi2b transcript or other genes related to cancer measured in tumor samples Blood-based biomarkers, which may include serum cytokines, circulating immune cells, and circulating tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Brad Sumrow, MD, Study Director — Mersana Therapeutics
Locations (1):
- START Midwest, Grand Rapids, Michigan, United States